CLINICAL TRIAL: NCT03806673
Title: Is There a Relation Between Unilateral Epidural Block and Repeated Epidural Anesthesia?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Ain Shams Un
Record Dates: First submitted 2019-01-12; First posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Incidence; Unilateral; Epidural Block
Keywords: unilateral, ,; epidural block; repeated epidural
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: double blinded randomized
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primipara (Active Comparator): primipara subjected to their first epidural block
  Interventions: Drug: marcaine
- multipara (Active Comparator): multipara subjected to their repeated epidural block.
  Interventions: Drug: marcaine

INTERVENTIONS:
Drug: marcaine — epidural block

SUMMARY:
epidural block is today the most common method of pain relief during labor. With increased use of epidural analgesia, many women are found in the second or third pregnancy and require repeated epidural analgesia. But there was a higher incidence of unilateral blockade among women receiving their repeated epidural which causes patient unsatisfaction.

Objectives: Examination of the performance and outcome of women receiving their first versus repeated epidural block.

Patients and methods: The study included 140 American Society of Anesthesiologists (ASA) Physical Status II patients (age range 20 to 40 years) and scheduled for normal vaginal delivery. The patients were divided randomly into two equal groups. Group (A) in which 70 women primipara subjected to their first epidural block while group (B) in which 70 women multipara subjected to their repeated epidural block. For each patient, the following data were collected: demographic data, details of labor (gestation, cervical dilatation), visual analogue scale (VAS) before the epidural and 30 minutes after injection of local anesthetic and incidence of unilateral block.

DETAILED DESCRIPTION:
This study was performed after obtaining approval from the ethical committee of the Ain Shams University. Sample of 140 healthy ASA II female patients, 20-40 years of age, scheduled for normal vaginal delivery. Patients were randomly allocated by computer-generated random number list into two study groups of 70 patients each.

Group (A) in which 70 primipara women subjected to their first epidural block while group (B) in which 70 multipara women subjected to their repeated epidural block. The study was carried out between January 2018 and March 2018.

Patients were excluded for:

* Any physical reason for difficult epidural performance e.g.: morbid obesity, or scoliosis,
* Severe hypertension,
* Congestive heart failure,
* Coagulopathy,
* Significant hepatic or renal disease,
* Or withdrawal of consent. All patients in this study were subjected to a detailed pre-anesthetic evaluation. All basic investigations according to the hospital protocol (e.g. serum hemoglobin, platelet count, coagulation profile) were checked.

The patient's demographic data, details of labor (gestation, cervical dilatation), details of epidural insertion were recorded by the anesthetist performing the epidural.

The patient was asked to mark a visual analogue scale (VAS) (figure 1) before the epidural and 30 minutes after injection of local anesthetic. Also incidence of unilateral epidural block is reported 30 minutes after injection of local anesthetic.

Figure (1): Visual analog scale 2.2 Anesthetic technique On arrival to operation room; 18 g cannula was inserted then 500 ml of Ringer solution was infused while performing the epidural.

Basic monitors including automatic blood pressure measurements, five lead ECG monitor, and finger pulse oximetry were applied to all patients.

A standard procedure was followed for epidural insertion and establishment of block. With the patient in the sitting position the midline approach was used using 16-g Tuohy needle and the epidural space was identified by loss of resistance to air, as is our routine practice.

Once the epidural space was reached, Bupivacaine 0.25% plain, was given in three 5 ml increments at five-minute intervals, the first administered through the needle while the patient is in sitting position, and then through the catheter with the patient in supine position.

Multi-orifice catheters were inserted and fixed to a standard 4 cm extra to the distance between the skin and epidural space. At the time of insertion of the catheter the patient was asked to report any pain or tingling experienced.

The operator recorded the ease of insertion of the catheter (difficult or easy) and the occurrence of blood in needle or catheter. Epidurals were performed by the same anesthetists.

At 30 min after injection of bupivacaine, the second VAS was completed and the level of blockade checked by cold sensation test. If an inadequate level was noted (less than T10), the pain score remained high or increased, or the patient complained of poor pain relief she was asked to describe the site and type of pain experienced.

A unilateral block was defined as the description by the patient of worse pain on one side than the other, or pain on one side only, combined with either a 30-min pain score minimally changed or increased from time zero or a low level of blockade on the painful side, or both. If unilateral or inadequate block occurred the catheter was withdrawn 0.5-1 cm and a further 5 ml bupivacaine 0.25% was administered with the patient lying on the unblocked side. If the block was still inadequate, epidural fentanyl 50 microgram was given and if still inadequate the catheter was removed and a second epidural catheter inserted in another interspace.

The number of repeat injections of bupivacaine and length of time between epidural insertion and delivery were noted, as well details of previous epidurals in the multiparous women.

Sample size estimation:

To show a difference in the incidence of unilateral block between the two groups with p-value < 0.05 and power 80%, we needed at least 60 patients per group.

Statistical analysis:

Analysis of data was done by IBM computer using SPSS (statistical program for social science, version 16) as follows:

* Description of quantitative variables as mean ± SD.
* Description of quantitative variables as number and percentage. Statistical analysis was performed using statistical tests included Student's t-test, Chi square test and table analysis. P value <0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* healthy ASA II female patients,

  * 20-40 years of age,
  * scheduled for normal vaginal delivery.
  * Exclusion Criteria:
* - Any physical reason for difficult epidural performance e.g.: morbid obesity, or scoliosis,
* Severe hypertension,
* Congestive heart failure,
* Coagulopathy,
* Significant hepatic or renal disease,
* Or withdrawal of consent.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 140 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
sensation | 30 minutes after injection of local anesthetic
  by cold skin test

CONTACTS AND LOCATIONS:
Locations (1):
- Ramymahrose, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No